CLINICAL TRIAL: NCT07166146
Title: Timing and Outcomes of Recovery After intraCerebral Hemorrhage
Acronym: TORCH
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: Hongtao TORCH
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Intracerebral Haemorrhage; Intracerebral Hemorrhage
Keywords: Intracerebral Haemorrhage; Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surgical interventions — By leveraging a wide array of surgical interventions - including endoscopic surgery, minimally invasive surgery combined with urokinase, and craniotomy - the TORCH registry intends to provide a granular view of early hematoma evacuation surgical interventions and their impact on patient recovery and quality of life.

SUMMARY:
The TORCH registry is a prospective, observational cohort study, which will collect detailed, longitudinal data on the clinical characteristics, treatment modalities, and outcomes of patients with ICH. By leveraging a wide array of surgical interventions - including endoscopic surgery, minimally invasive surgery combined with urokinase, and craniotomy - the TORCH registry intends to provide a granular view of early hematoma evacuation surgical interventions and their impact on patient recovery and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subject Age is ≥18 to ≤80 years
* Subject with a Head CT/CTA that demonstrates an acute, spontaneous, primary, supratentorial ICH, assessed via standard of care techniques
* Subject recieving a surgery intervention
* Subject has a NIHSS score ≥ 6 or GCS score 5≤GCS≤15
* Subject has a baseline Modified Rankin Scale (mRS) Score ≤ 1

Exclusion Criteria:

* Secondary intracerebral hemorrhage (with leading cause, e.g., Moyamoya disease, arteriovenous malformation, intracranial aneurysm, tumor, brain trauma)
* Pre-stroke life expectancy < 1 year for severe comorbidities (e.g., Progressive malignant tumor, severe chronic heart failure [NYHA: III-IV], severe chronic obstructive pulmonary disease [III-IV], chronic kidney disease requiring hemodialysis)
* Patients with platelet count < 100,000, INR > 1.4, or an elevated PT or APTT (reversal of coumadin is permitted but the patient must not require coumadin during the acute hospitalization). Irreversible coagulopathy either due to medical condition or prior to randomization
* Pregnant (positive pregnancy test) or lactating females (likelihood of altered coagulation function associated with the high estrogen/progesterone state)
* Irreversibly impaired brainstem function (bilateral fixed, dilated pupils and extensor motor posturing), GCS less than or equal to 4

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Functional Outcome | 6 months after onset
  modified Rankin Score (mRS) 0=no symptoms, 1=no significant disability, 2=slight disability, 3= moderate disability, 4=moderate severe disability, 5=severe disability, 6=death

SECONDARY OUTCOMES:
Functional Outcome | 3 months after onset
  modified Rankin Score (mRS) 0=no symptoms, 1=no significant disability, 2=slight disability, 3= moderate disability, 4=moderate severe disability, 5=severe disability, 6=death
Safety - Procedure -Related Mortality | 30 days after onset
  Safety will be assessed by determining procedure-related mortality by comparing rates of mortality at 30 days
EQ-5D-5L | 6 months after onset
  EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. EQ-5D-5L
Functional Status in Daily Life | 6 months after onset
  180±14 days of Barthel index

CONTACTS AND LOCATIONS:
Locations (1):
- The Department of Neurosurgery, China International Neuroscience Institute, Xuanwu Hospital, Capital Medical University,, Beijing, China